CLINICAL TRIAL: NCT05475392
Title: Effects of Stretching Exercises With and Without Post Isometric Relaxation on Neck Pain and Muscular Spasm in Breastfeeding Women
Brief Title: Effects of Post Isometric Relaxation With and Without Stretching Exercises on Neck Pain and Muscle Spasm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/22/0523
Record Dates: First submitted 2022-07-24; First posted 2022-07-26 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Neck Pain; Muscle Spasm
Keywords: Breastfeeding women; Muscle spasm; Neck pain; Post Isometric Relaxation; Stretching
MeSH Terms: conditions — Neck Pain; Spasm

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stretching Exercise with PIR on neck pain and muscle spasm in breastfeeding women (Experimental): Experimental Group (Group A) will receive stretching with Post Isometric Relaxation and conventional treatment. Treatment will be given for five days per week for total two weeks. Pain will be assessed through VAS scale and MJM scale will be used to assess spasm. Assessment was done 2 times pretreatment and post treatment.
  Interventions: Other: Traditional Physical Therapy; Other: Post Isometric Relaxation
- Stretching Exercise without PIR on neck pain and muscle spasm in breastfeeding women (Active Comparator): Active Compatitor (Group B) will receive only stretching and conventional treatment. Treatment will be given for five days per week for total two weeks. Pain will be assessed through VAS scale and MJM scale will be used to assess spasm. Assessment was done 2 times pretreatment and post treatment.
  Interventions: Other: Traditional Physical Therapy

INTERVENTIONS:
Other: Traditional Physical Therapy — A 2-week physical therapy program will be arranged. Each patient will be given 60 min session , 10 min for neck ROMS (10 reps for each ROM) , 10 min neck Isometrics (5 reps on each side) , 30 sec static gentle stretch of levator scapulae (3reps) , 30 sec static gentle stretch of trapezius (3reps), 5 min Soft tissue manipulation , 5 min Shoulder shrugging (10reps) , 10 min for PIR
Other: Post Isometric Relaxation — The exercise will be combined with the baseline treatment 3 sets PIR will be applied per session.The hypertonic muscle is taken to a length just short of pain, or to the point where resistance to movement is first noted. A submaximal (10-20%) contraction of the hypertonic muscle is performed away from the barrier for between 5 and 10 seconds and the therapist applies resistance in the opposite direction. The patient should inhale during this effort. After the isometric contraction, the patient is asked to relax and exhale while doing so. Following this, a gentle stretch is applied to take up the slack till the new barrier. Starting from this new barrier, the procedure is repeated two or three times.
  Arms: Stretching Exercise with PIR on neck pain and muscle spasm in breastfeeding women

SUMMARY:
Neck pain is common in the adult general population, disabling and costly Lifetime, which constituted a great problem facing the mother during breast feeding period. The studies showed that poor knowledge and wrong position for breastfeeding influence their own health as well as baby's health. Stretching exercises are one of the manual physical therapy methods that can be used in the treatment of mechanical neck pain) Muscle energy techniques (MET) were originally developed to treat soft tissue, mobilize joints, stretch tight muscles and fascia, reduce pain and to improve circulation and lymphatic drainage. This study aims at applying stretching along with MET technique (post isometric relaxation) to see the combined effect of these two techniques and comparing that group with another one that is only applied stretching and baseline treatment. A randomized clinical trial will be undertaken. Non probability convenient sampling will be used. Forty-six patients with neck pain and muscular spasm will be randomly allocated. Twenty-three participants will be allocated with lottery method in each group. The former group will receive Stretching with MET (post isometric relaxation), and the latter group will receive static stretching only. Both groups will also receive baseline therapy. Treatment will be given once a day daily for 14 days. A visual analogue scale (VAS) will be used to measure the intensity of pain and MMJ questionnaire for muscular spasm. Data will be collected before and at the end of treatment at the 14th day. To analyze data SPSS version 29 will be used.

DETAILED DESCRIPTION:
Neck pain is common in the adult general population, disabling and costly Lifetime, which constituted a great problem facing the mother during breast feeding period. The studies showed that poor knowledge and wrong position for breastfeeding influence their own health as well as baby's health. Stretching exercises are one of the manual physical therapy methods that can be used in the treatment of mechanical neck pain) Muscle energy techniques (MET) were originally developed to treat soft tissue, mobilize joints, stretch tight muscles and fascia, reduce pain and to improve circulation and lymphatic drainage. This study aims at applying stretching along with MET technique (post isometric relaxation) to see the combined effect of these two techniques and comparing that group with another one that is only applied stretching and baseline treatment. A randomized clinical trial will be undertaken. Non probability convenient sampling will be used. Forty-six patients with neck pain and muscular spasm will be randomly allocated. Twenty-three participants will be allocated with lottery method in each group. The former group will receive Stretching with MET (post isometric relaxation), and the latter group will receive static stretching only. Both groups will also receive baseline therapy. Treatment will be given once a day daily for 14 days. A visual analogue scale (VAS) will be used to measure the intensity of pain and MMJ questionnaire for muscular spasm. Data will be collected before and at the end of treatment at the 14th day. To analyze data SPSS version 29 will be used.

ELIGIBILITY:
Inclusion Criteria:

* Women of age from 25 to 35years,
* All patients must be in breastfeeding period at least 6 weeks after delivery,
* BMI of women must be less than 30 kg/m²,
* Parity of women must not more than 3 times

Exclusion Criteria:

* Patient should not be in Pregnancy phase.
* There should not be Positive neurological examination
* Cervical spine surgery or stenosis patients should not be included
* Metastases patients should not be included.
* Participants should not have aassociated pathology of the upper cervical region or upper limb that may cause overlapping with the clinical finding as referred pain from costotransverse joint, rotator cuff tendonitis, and cervical rib syndrome

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Breast Feeding Women
Enrollment: 46 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-01-08 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
VAS (Visual Analogue Scale) | 2 Weeks
  For Neck pain. VAS will be described to patients using a 100 mm horizontal line with 0 representing "no pain" and 10 representing "worst pain imaginable". Patient marked a point on the line that matched the current amount of the pain he or she felt.
MMJ questionnaire (Muscle and Joint Measure) | 2 Weeks
  For muscular spasm.The MJM has potential research and clinical value for addressing the musculoskeletal symptoms. Readings with 0 to 10 on it. 0 represents to no muscle cramps or spasm at all and 10 represents to cramps and spasms as bad as they can possibly be.

CONTACTS AND LOCATIONS:
Overall Officials: Sabiha Arshad, M.Phil, Principal Investigator — Riphah International University
Locations (1):
- Jinnah Hospital , Gynea Ward, Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ojukwu CP, Okpoko CG, Ikele IT, Ilo IJ, Ede SS, Anekwu NE, Okemuo AJ, Anekwu EM, Ugwu SU, Ikele CN. Neck Muscles' Responses to Cradle, Cross-cradle and Football Breastfeeding Hold Positions in Nursing Mothers: A Preliminary Study. Niger J Clin Pract. 2022 May;25(5):563-568. doi: 10.4103/njcp.njcp_630_20. PMID 35593596
- [Background] Rani S, Habiba UE, Qazi WA, Tassadaq N. Association of breast feeding positioning with musculoskeletal pain in post partum mothers of Rawalpindi and Islamabad. J Pak Med Assoc. 2019 Apr;69(4):564-566. PMID 31000863
- [Background] Romanowski MW, Spiritovic M, Romanowski W, Straburzynska-Lupa A. Manual Therapy (Postisometric Relaxation and Joint Mobilization) in Knee Pain and Function Experienced by Patients with Rheumatoid Arthritis: A Randomized Clinical Pilot Study. Evid Based Complement Alternat Med. 2020 Aug 19;2020:1452579. doi: 10.1155/2020/1452579. eCollection 2020. PMID 32922504
- [Background] Lewit K, Simons DG. Myofascial pain: relief by post-isometric relaxation. Arch Phys Med Rehabil. 1984 Aug;65(8):452-6. PMID 6466075